CLINICAL TRIAL: NCT07128264
Title: The Effect of Laughter Yoga on Patients With Ankylosing Spondylitis: A Randomized Controlled Trial
Brief Title: The Effect of Laughter Yoga on Patients With Ankylosing Spondylitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, SELANAY ÜNAL, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU-SBE-SU-01
Record Dates: First submitted 2025-08-12; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Ankylosing Spondylitis (AS)
Keywords: Ankylosing spondylitis(AS),Nursing,Pain,Depression/anxiety/stress,Laughter yoga
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Two groups with a laughter yoga control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Patients in the intervention group will be divided into 2 groups of 15 people. A total of 12 sessions of laughter yoga will be applied to the intervention group in the form of meetings via the Microsoft teams application, in 45-minute sessions 2 times a week for 6 weeks. Laughter yoga sessions will be held every week on ………. and ………. days. The days of the laughter yoga program will be decided in accordance with the patients, together with the participating patients, on the basis of research. Before the laughter yoga, an informative message will be sent to each patient in the intervention group about the meeting and the patients' participation in the sessions will be checked with a follow-up chart.
  Interventions: Behavioral: Laughter Yoga
- Control (No Intervention): Laughter yoga will not be applied to patients in the control group.

INTERVENTIONS:
Behavioral: Laughter Yoga — Laughter eliminates feelings such as hopelessness, anger, and anxiety, thereby alleviating stress, depression, and anxiety, raising the pain threshold, reducing stress, accelerating blood circulation, strengthening immunity, improving quality of life, strengthening memory, reducing tension, and relaxing muscles. Based on these positive effects, laughter yoga is a complementary treatment method that combines humor and laughter. Laughter yoga sessions will be conducted online via Microsoft Teams in a quiet and peaceful environment at home.
  The first 10-minute section consists of warm-up exercises (warming up and clapping). The second 10-minute section consists of deep breathing exercises that prepare the lungs for laughter. The third 10-minute section consists of childlike games that induce laughter without humor. The fourth and final 15-minute section consists of laughter exercises that enable laughter without any jokes, comedy, or humor.
  Arms: Intervention

SUMMARY:
This study will be conducted to evaluate the effects of laughter yoga on disease activity, pain, functional status, depression/anxiety/stress, and quality of life in ankylosing spondylitis patients.

DETAILED DESCRIPTION:
Ankylosing spondylitis is a common inflammatory rheumatic disease that primarily affects the axial skeleton, causes characteristic inflammatory back pain, and can lead to progressive structural and functional impairments and a decrease in quality of life.

The main symptoms of the disease include severe back pain and spinal stiffness, as well as inflammation of the peripheral joints, hips, and fingers/toes. In advanced cases, inflammation of the spinal joints may lead to fusion of the spine and associated functional limitations. Research has shown that physical symptoms in AS patients are accompanied by psychological symptoms such as fatigue, stress, depression, and anxiety. All of these factors can lead to a deterioration in quality of life.

Material and Method: This randomized controlled trial will be conducted with a total of 60 patients (30 intervention and 30 control) who agreed to participate in the study and visited the Rheumatology Outpatient Clinic at Erzurum City Hospital. Patients in the intervention group will undergo laughter yoga sessions twice a week for 45 minutes over a period of 6 weeks. Patient information forms will be used to collect research data, and the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) will be used as the primary measurement tool. Secondary measurement tools will include the Visual Analogue Scale (VAS) Pain Scale, Bath Ankylosing Spondylitis Functional Index (BASFI), Depression/Anxiety/Stress Scale (DASS-42), and Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL).

Application of the research: Patients visiting the outpatient clinic will be informed about the study, and written consent will be obtained from patients who agree to participate in the study. Inclusion criteria for the study will be evaluated. Patients will be administered the patient information form, Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Visual Analogue Scale (VAS), Bath Ankylosing Spondylitis Functional Index (BASFI), DASS-42, and Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) scales. Patients will be assigned to the intervention and control groups according to the randomization list.

Intervention group:

The researcher will provide general information about laughter yoga to each patient in the intervention group, and the Microsoft Teams application will be installed on the patients' smartphones for the laughter yoga sessions. Patients' phone numbers will be collected for communication, and WhatsApp groups will be created to facilitate communication. The days of the laughter yoga program will be decided in consultation with the patients participating in the study, taking into account the patients' schedules. Prior to laughter yoga, each patient in the intervention group will receive an informational message about the meeting, and patients' attendance at the sessions will be monitored using a tracking chart.

Patients in the intervention group will be divided into two groups of 15. The intervention group will undergo a total of 12 laughter yoga sessions over 6 weeks, with two 45-minute sessions per week via Microsoft Teams. Laughter yoga sessions will be held every week on ………. and ………. days.

Laughter yoga will not be applied to patients in the control group. At the end of the 6th week, patients in both groups will come to the rheumatology outpatient clinic and final test measurements will be taken. At the outpatient clinic, patients will be administered the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Vas Pain Scale, Bath Ankylosing Spondylitis Functional Index (BASFI), Depression/Anxiety/Stress Scale (DASS-42), and Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) will be administered to patients at the outpatient clinic.

For patients in the intervention group, final test measurements will be conducted at least two days after the session to exclude the acute effects of laughter yoga.

Patients in both the intervention and control groups will continue their routine treatments for six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Those diagnosed with ankylosing spondylitis,
* Those who scored 10 or above on the depression scale, 8 or above on the anxiety scale, and 15 or above on the stress scale of the Depression-Anxiety-Stress Scale
* Are over 18 years of age,
* Have no hearing or communication problems,
* Possess a smartphone,
* Have no physical problems that would prevent them from performing yoga exercises (bleeding hemorrhoids, any type of hernia, persistent cough, incontinence, hypertension, major psychiatric disorders, pregnancy, flu, epilepsy, or surgery within the last 3 months, etc.)
* Ankylosing spondylitis patients who volunteer to participate in the study will be included in the study sample.

Exclusion Criteria:

* Patients who do not participate in laughter yoga
* Patients who wish to withdraw from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-29 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) | 6 weeks
  BASDAI, which assesses disease activity in ankylosing spondylitis, was developed by Garret and colleagues in 1994 . The scale includes six questions to assess disease activity over the past week, consisting of fatigue, spinal pain, joint swelling, tenderness, and morning stiffness. The patient's symptoms are scored on a scale of 0 to 10 (0 = none, 10 = very severe). When calculating the total score, the average of questions 5 and 6 is added to the scores of questions 1, 2, 3, and 4, and the total is divided by 5 to determine the total score. The total score of the scale ranges from 0 to 10. Higher scores indicate greater disease activity.

SECONDARY OUTCOMES:
Pain Scale (Visual Analog Scale) | 6 weeks
  The VAS is a straight line used to measure the variability of pain and indicates the continuity of pain. At one end of this line is painlessness (0), and at the other end is the most severe pain (10) that can occur.
Bath Ankylosing Spondylitis Functional Index (BASFI) | 6 weeks
  The BASFI, which assesses functional status in ankylosing spondylitis, was developed in 1994 by Calin et al. The scale assesses patients' ability to put on socks/tights, bend forward from the waist, reach high, get up from a chair or the floor without support, stand without support, look sideways over their shoulders without turning their body, climbing stairs without assistance, performing activities requiring physical strength, and performing activities at home/work. Eight of the questions in the scale relate to daily living activities, and two relate to coping with life. Patients are asked to rate how much difficulty they experience while performing each activity on a visual analog scale from 0 to 10 (0 = easy, 10 = impossible). The scale is scored by summing the points given for each question and dividing by 10 to obtain the average. The total score ranges from 0 to 10. An increase in the BASFI score is interpreted as a decrease in functional capacity.
DASS-42 Scale (Depression-Anxiety-Stress Scale) | 6 weeks
  The scale is a 4-point Likert scale consisting of 3 subscales (depression,anxiety, stress).Each subscale has 14 items,for a total of 42 items on the scale.The depression items assess feelings of helplessness,worthlessness, dissatisfaction,loss of interest,and low energy levels.Anxiety items measure muscle response levels,the individual's autonomic arousal,and subjective and situational anxiety.Stress items assess discomfort,difficulty relaxing, overreaction,nervous arousal,intolerance,easy sadness,and boredom levels. Depression is categorized as remission(0-9),mild(10-13),moderate(14-20),severe (21-27),and very severe (28-42);anxiety is categorized as remission (0-7),mild (8-9),moderate (10-14),severe (15-19),and very severe(20-42);and stress remission (0-14),mild(15-18),moderate(19-25),severe(26-33),and very severe (34-42)into five categories.Each of the depression,anxiety,and stress scores ranges from 0 to 42,and as the score increases,depression,anxiety,and stres also increases.
Ankylosing Spondylitis Quality of Life Questionnaire (ASQoL) | 6 weeks
  The Ankylosing Spondylitis Quality of Life Questionnaire was developed in 2007 by Doward and colleagues to assess the quality of life of patients with this specific disease. The questionnaire consists of 18 items related to the symptoms, functioning, and concerns associated with the disease. Each statement is followed by "no" and "yes" options. Each 'yes' answer is scored as one point, while each "no" answer is scored as zero points. The total score of the scale ranges from 0 to 18. An increase in the total score indicates a lower quality of life for the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Emine KIYAK, Prof.Dr., Study Director — Ataturk University

IPD SHARING:
Plan to Share IPD: No